CLINICAL TRIAL: NCT00768235
Title: Influence of Yoga Program in Respiratory Function of Older Women
Brief Title: Yoga Program in Respiratory Function
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Catholic University of Brasília (Other)
Responsible Party: Lidia Mara Aguiar Bezerra
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCByoga123; UCByoga12345
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Elderly
Keywords: Sedentary elderly women that had medical assignment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: yoga group (Experimental): Yoga group
  Interventions: Other: yoga practice
- 2: control group (No Intervention)

INTERVENTIONS:
Other: yoga practice — The yoga program comprised 70 min sessions, 3 times/week during 12 weeks
  Arms: 1: yoga group

SUMMARY:
This study tested the hypothesis that yoga practice can improve respiratory function in the elderly.

DETAILED DESCRIPTION:
Maximal inspiratory and expiratory pressure (IPmax and EPmax) were assessed by a manovacuometer and tidal volume (VT), vital capacity (VC) and minute ventilation (VE) were assessed by a ventilometer. The yoga program comprised 70 min sessions, 3 times/week during 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary women

Exclusion Criteria:

* Physical impairment

Ages: 51 Years to 76 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-03; Primary Completion 2007-03 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory and expiratory pressure (IPmax and EPmax) were assessed by a manovacuometer and tidal volume (VT), vital capacity (VC) and minute ventilation (VE) were assessed by a ventilometer | pre-intervention and post-intervention

SECONDARY OUTCOMES:
Maximal inspiratory and expiratory pressure (IPmax and EPmax) were assessed by a manovacuometer and tidal volume (VT), vital capacity (VC) and minute ventilation (VE) were assessed by a ventilometer | pre-intervention and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Lidia MA Bezerra, Ms., Principal Investigator — catholic University of Brasilia
Locations (1):
- Catholic university of brasilia, Brasília, Federal District, Brazil

REFERENCES:
- [Background] Buchman AS, Boyle PA, Wilson RS, Leurgans S, Shah RC, Bennett DA. Respiratory muscle strength predicts decline in mobility in older persons. Neuroepidemiology. 2008;31(3):174-80. doi: 10.1159/000154930. Epub 2008 Sep 11. PMID 18784416
- See also: article — http://www.ncbi.nlm.nih.gov/pubmed/18784416?ordinalpos=1&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum